CLINICAL TRIAL: NCT03653676
Title: The Pro-Inflammatory Effects of Acute Exercise in Children With Sickle Cell Anemia
Brief Title: Sickle Cell Pro-Inflammatory Response to Interval Training Study
Acronym: SPRINTS
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: University of Illinois at Chicago (Other); St. Jude Children's Research Hospital (Other); Columbia University (Other); University of California, Irvine (Other)
Responsible Party: Principal Investigator, Robert I. Liem, Principal Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2017-881
Record Dates: First submitted 2018-01-02; First posted 2018-08-31 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Anemia; Sickle Cell Disease; Exercise; Fitness; Asthma; Inflammation
MeSH Terms: conditions — Anemia, Sickle Cell; Motor Activity; Asthma; Inflammation | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — In this study, blood specimens will be collected at baseline and as part of pre and post CIIT exercise challenge. These studies will include routine clinical tests as well as biomarkers of inflammation and cellular adhesion. In a subset of participants at Lurie Children's, samples for genomic studies will be collected pre and post CIIT exercise challenge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with SCA: Children and adolescents with SCA confirmed by hemoglobin analysis randomized to either moderate or vigorous intensity exercise test (CIIT)
  Interventions: Other: Exercise Test (CIIT)
- Controls without SCA: Children and adolescents without SCA or sickle cell trait randomized to either moderate or vigorous intensity exercise test (CIIT)
  Interventions: Other: Exercise Test (CIIT)

INTERVENTIONS:
Other: Exercise Test (CIIT) — The CIIT exercise test will consist of 8 bouts (2 minute each) of constant workload cycling with rest periods (1 minute each) in between each bout of exercise. Subjects and controls will be randomized to either a moderate intensity or vigorous intensity, defined as 50% or 70% of the maximal workload achieved on the maximal cardiopulmonary exercise test (CPET).

SUMMARY:
Recommendations for exercise prescription currently do not exist for individuals with sickle cell anemia (SCA) despite the known impact that SCA-related complications has on physical functioning and fitness. A major barrier to increasing physical activity in SCA is the concern that the well-described inflammatory effects of exercise could precipitate or exacerbate complications such as vaso-occlusive pain or airway bronchoconstriction (i.e. exercise-induced asthma). Although the investigator's preliminary data suggest that increasing physical activity may be beneficial rather than harmful in children with SCA, the pro-inflammatory effects associated with repeated bouts of moderate to vigorous exercise remain poorly understood in this population. The long term goal is to address the safety and health impact of regular exercise in children with SCA. This proposal would help establish the safety of moderate to vigorous intensity exercise in children with SCA and importantly, will inform the design of future clinical trials focused on exercise training as a transformative strategy to improve fitness and overall well-being in this population.

DETAILED DESCRIPTION:
The investigator's plan to evaluate the effect of acute exercise and exercise intensity on circulating systemic pro-inflammatory mediators and airway bronchoconstriction in SCA. The investigators hypothesize that regular exercise at moderate to vigorous intensity is safe for children with SCA and do not precipitate SCA-related symptoms. In this multicenter study, 70 non-asthmatic children with SCA and 70 controls without SCA will first undergo a maximal cardiopulmonary exercise test (CPET), then be randomized to an exercise challenge by controlled intensity interval training (CIIT) at either moderate or vigorous intensity (8 exercise bouts at 50% or 70% peak workload, respectively). The Investigator's Aims are to: 1) Determine the influence of exercise intensity on the acute inflammatory response to exercise, defined by an increase in soluble vascular cell adhesion molecule (VCAM) and other adhesion molecules, and 2) Define the effect of moderate to vigorous exercise on forced expiratory volume in 1 second (FEV1) and acute bronchoconstriction in children with SCA. The investigators will also explore exercise- induced changes in gene and microRNA expression in peripheral blood mononuclear cells, tissue oxygenation during exercise by near infrared spectroscopy as well as the role of hyperventilation in bronchoconstriction using eucapnic voluntary hyperventilation testing in a subset of participants.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female, aged 10 years to 21 years old
* Diagnosis of hemoglobin SS or S/Beta0 thalassemia confirmed by hemoglobin electrophoresis

Exclusion Criteria:

* Inability to perform CPET due to physical limitation (e.g. severe hip osteonecrosis or stroke)
* Enrollment on chronic transfusion program
* History of exercise-induced arrhythmia or syncope
* Diagnosis of asthma, defined as physician diagnosis or use of daily asthma medications
* Known exercise-induced bronchoconstriction, defined as physician diagnosis by exercise challenge test
* History of any cardiac diagnosis precluding exercise testing, unless cleared by a cardiologist
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study will plan to enroll a total of 70 non-asthmatic subjects with SCA and 70 controls without SCA across all sites. Male or female, aged 10 years to 21 years old. Diagnosis of hemoglobin SS or S/Beta0 thalassemia confirmed by hemoglobin electrophoresis.
  Children and young adults on hydroxyurea are eligible but must be at steady state at time of enrollment, defined as stable dosing for at least 2 months, without anticipated changes in dose during study participation.
  Race and age-matched controls without SCA or sickle cell trait will be recruited among friends, relatives, siblings or individuals from similar communities to minimize confounding socio-demographic variables that may impact baseline fitness. Controls will be required to be 10 through 21 years of age.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Biomarker- VCAM-1 | Through study completion, approximately 2 years
  Change in soluble vascular cell adhesion molecule VCAM-1 in ng/mL

SECONDARY OUTCOMES:
Biomarker - ICAM-1 | Through study completion, approximately 2 years
  Change in intercellular adhesion molecule-1 in ng/mL
Biomarker - PECAM-1 | Through study completion, approximately 2 years
  Change in platelet endothelial cell adhesion molecule-1 in ng/mL
Biomarker - L-selectin | Through study completion, approximately 2 years
  Change in L-selectin in ng/mL
Biomarker - E-selectin | Through study completion, approximately 2 years
  Change in E-selectin in ng/mL
Biomarker - P-selectin | Through study completion, approximately 2 years
  Change in P-selectin in ng/mL
Biomarker - IL-6 | Through study completion, approximately 2 years
  Change in interleukin-6 in pg/mL
Exercise spirometry | Through study completion, approximately 2 years
  Forced expiratory volume in 1 second (FEV1 mesured in % of normal predicted value)
Near infrared spectroscopy (NIRS) - total oxygen saturation | Through study completion, approximately 2 years
  Near infrared spectroscopy (NIRS) derived measurements (total oxygen saturation (StO2) in the pre-frontal cortex and vastus lateralis muscle) in %
Near infrared spectroscopy (NIRS) - oxygenated hemoglobin | Through study completion, approximately 2 years
  Near infrared spectroscopy (NIRS) derived measurements (oxygenated hemoglobin in the pre-frontal cortex and vastus lateralis muscle) in %
Near infrared spectroscopy (NIRS) - deoxygenated hemoglobin | Through study completion, approximately 2 years
  Near infrared spectroscopy (NIRS) derived measurements (deoxygenated hemoglobin in the pre-frontal cortex and vastus lateralis muscle) in %
Genomic studies | Through study completion, approximately 2 years
  Gene and microRNA expression in mononuclear cells measured by fold change
Asthma risk screening - ISAAC questionnaire | Through study completion, approximately 2 years
  International Study of Asthma and Allergies in Childhood (ISAAC) screening questionnaire for rhinitis and eczema based on yes/no responses and point system to determine severity of condition (e.g. for rhinitis, 0 to 3 points (most severe); for eczema, 0 to 4 points (most severe)).
Asthma risk screening - FeNO measurement | Through study completion, approximately 2 years
  Exhaled nitric oxide (FeNO) in ppb)
Asthma risk screening - Urinary Leukotrienes | Through study completion, approximately 2 years
  Urine leukotriene (LTE4) in pg/mg)
Eucapnic voluntary hyperventilation (EVH) spirometry | Through study completion, approximately 2 years
  Forced expiratory volume in 1 second (FEV1 in % of normal predicted value) will be taken after EVH at 5, 10, 15, and 30 minutes to assess exercise induced bronchoconstriction in a subset of participants.
Adverse events | Through study completion, approximately 2 years
  Safety outcomes including number of cardiopulmonary complications, vaso-occlusive pain or other adverse events related to exercise and EVH reported as incidence (number and %).
Patient reported physical functioning - fatigue | Through study completion, approximately 2 years
  NIH PROMIS questionnaire for fatigue using appropriate raw summed and T scores with higher scores indicating worse fatigue (pediatric - raw 0 to 40, T score 30.3 to 84; parent proxy - raw 0 to 40, T score 34 to 85; adult - raw 8 to 40, T score 33.1 to 77.8)
Patient reported physical functioning - mobility | Through study completion, approximately 2 years
  NIH PROMIS questionnaire for mobility using appropriate raw summed, scale or T scores with higher scores indicating better mobility (pediatric - raw 0 to 32, T-score 15.2 to 58.5; adult - raw 8 to 40, T-score 20.9 to 59.7; parent proxy - raw 0 to 32, scale 14 to 56)
Patient reported physical activity level | Through study completion, approximately 2 years
  NHANES physical activity questionnaire for frequency of moderate versus vigorous physical activity in number of days in typical week (range 0 to 7 days with higher number indicating more days spent in moderate or vigorous activity) and time spent in typical day (0 to > 2 hours with higher number indicating more hours spent in moderate or vigorous activity)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Liem, MD, Principal Investigator — Ann and Robert H. Lurie Childrens Hospital
Locations (3):
- United States (3):
  - University of Illinois at Chicago, Chicago, Illinois
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cohen RT, Hankins JS, Ness KK, Hsu LL, Baynard T, Tang A, Radom-Aizik S, Guerrero K, Rodeghier M, Liem RI. Acute Exercise Challenge and Airway Dynamics in Youth With Sickle Cell Anemia: A Multicenter Study. Am J Hematol. 2025 Dec 20. doi: 10.1002/ajh.70170. Online ahead of print. PMID 41422377